CLINICAL TRIAL: NCT07151521
Title: Application Value of Novel PET Tracers Targeting CAF in ANCA-Associated Vasculitis
Brief Title: (68)Ga-FAPI PET/CT in Patients With ANCA-associated Vasculitis
Acronym: GFPIPWAAV
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-432
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: ANCA-associated Vasculitis
Keywords: ANCA-associated vasculitis; FAPI; PET/CT; ILD; Kidney
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ANCA-associated vasculitis with interstitial lung disease
- ANCA-associated vasculitis without interstitial lung disease
- ANCA-associated vasculitis with renal dysfunction
- ANCA-associated vasculitis without renal dysfunction

SUMMARY:
Pulmonary and renal involvement are the most common clinical manifestations of antineutrophil cytoplasmic antibody(ANCA)-associated vasculitis (AAV). Studies have shown that both interstitial lung disease (ILD) and renal dysfunction are closely associated with poor prognosis in patients with AAV. Therefore, early identification of whether AAV patients have concomitant ILD and renal involvement is of great clinical importance for assessing disease severity, stratifying prognostic risk, and developing individualized treatment strategies.

Positron emission tomography (PET) is a noninvasive molecular imaging technique that can provide decision-making support for early and accurate diagnosis, timely intervention, as well as evaluation of treatment response and prognosis. In the same individual, PET enables whole-body localization of disease in a single examination, overcoming the limitation of conventional diagnostic methods that typically assess only one region at a time, thereby facilitating patient benefit.

In recent years, many novel PET tracers have been developed and introduced into clinical practice. 68Ga-Fibroblast Activation Protein Inhibitor (FAPI) has been studied in the diagnosis of various malignant and nonmalignant diseases; it targets fibroblast activation protein (FAP) and thus reflects the distribution of cancer-associated fibroblasts (CAFs). However, its clinical significance in AAV remains to be further investigated. This study aims to use a CAF-targeted novel PET tracer to conveniently and noninvasively detect the real-time distribution of lesions in patients, providing valuable information for personalized diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years;
2. Meeting the 2022 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria for ANCA-associated vasculitis;
3. Diagnosed with concomitant interstitial lung disease based on High-Resolution Computed Tomography (HRCT) images obtained within one year prior to enrollment, interpreted by two radiologists blinded to clinical information;
4. Complete clinical information available;
5. Signed and dated informed consent form;
6. Willingness to comply with the study procedures and cooperate throughout the entire study process.

Exclusion Criteria:

1. Presence of other rheumatic diseases;
2. Presence of other conditions that may cause interstitial lung disease or renal impairment, such as systemic lupus erythematosus, dermatomyositis, or rheumatoid arthritis;
3. History of, or planned, hematopoietic stem cell transplantation;
4. Presence of severe comorbidities deemed by the investigators to be unsuitable for participation in this clinical study, such as severe cardiopulmonary insufficiency, severe bone marrow suppression, or severe hepatic or renal insufficiency;
5. Acute abdominal emergencies such as intestinal perforation or complete intestinal obstruction;
6. Pregnant or potentially pregnant women, and lactating women;
7. Poor treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be recruited from Ruijin Hospital, Shanghai Jiao Tong University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease severity and activity in ANCA-associated vasculitis with concomitant interstitial lung disease and renal dysfunction as measured by 68Ga-FAPI PET/CT. | Within 4 weeks after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Ruiiin Hospital Shanghai JiaoTong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared because the informed consent obtained from participants did not include permission for public data sharing, and institutional as well as ethical guidelines require strict protection of participant confidentiality.